CLINICAL TRIAL: NCT01304849
Title: Phase II Study of Interim PET-CT Scan-guided Response Adapted Therapy in Hodgkin's Lymphoma
Brief Title: Use of Interim PET Scan to Modify Therapy in Advanced Hodgkin's Lymphoma in Order to Improve Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute WIA (Other)
Responsible Party: Principal Investigator, Prasanth Ganesan, Assistant Professor, Cancer Institute WIA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-HL-1
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; PET CT scan; Escalated BEACOPP; ABVD; Response adapted therapy
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primary (Experimental): Patients with aHL will receive 2 cycles of ABVD and undergo interim PET-2 scan- those with positive scans will receive 4 additional cycles of Esc BEACOPP while those with negative scans will receive 4 additional cycles of ABVD.
  Interventions: Drug: Escalated BEACOPP

INTERVENTIONS:
Drug: Escalated BEACOPP — Escalated BEACOPP chemotherapy will be delivered for those patients who are interim PET CT positive after 2 cycles of ABVD chemotherapy. The patients will receive 2-4 cycles of Escalated BEACOPP once in 3 weeks. The cycles will be delivered as follows:
  Bleomycin 10mg/m2 IV in day 8, Etoposide 200mg/m2 Day 1 to Day 3, Adriamycin 35mg/m2 on Day 1 IV, Cyclophosphamide 1200mg/m2 on Day 1 IV, Vincristine 1.4mg/m2 on Day 8 IV, Cap Procarbazine 100mg/m2 Day 1 to Day 7 PO, T Prednisolone 40mg D1-D7 of a 21 day cycle. With Inj Mesna 400mg/m2 0, 4 and 8 hours on the day of Cyclophosphamide Inj G-CSF will be started routinely from Day 9 till recovery of Absolute neutrophil counts ≥5000/cmm or Total WBC counts≥ 8000/cmm
  Other Names: EB

SUMMARY:
The current standard treatment for advanced Hodgkin's lymphoma 6-8 cycles of ABVD chemotherapy-this cures 70-80% patients. Those not cured after 8 cycles of ABVD have a poor outcome (<10% survival). More intensive chemotherapy like Escalated BEACOPP (EB) achieve higher cure rates have more side effects. Hence the investigators propose to use Interim PET CT scan (done after 2 cycles of ABVD) for early identification of poor responders (it is known that those with interim PET positive disease have a cure rate of less than 10-15% if continued with ABVD alone) and to use EB selectively in this population in an attempt to improve treatment outcomes - at the same time to limit side effects of therapy.

Thus, this study is an attempt to improve the outcome in the small subset of poor responders to ABVD chemotherapy by the early use of Escalated BEACOPP chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age 12-65 years old
* Newly diagnosed histology proven patients of advanced HL (stage IIb, III and IV)
* Patients' performance status ECOG 0-2
* Normal hematopoetic parameters except if due to marrow involvement by disease (WBC > 4000/cmm, Platelet count > 100,000/cmm)
* No uncontrolled hepatitis B/C infection; and normal LFT values with s -Bilirubin, SGOT and SGPT not more than 2.5 times upper limit of normal (unless initially due to liver involvement by disease)
* Serum Creatinine ≤ 2mg/dL unless elevated due to involvement by disease
* Cardiovascular/ Metabolic: No severe cardiac disease that would limit normal life expectancy or preclude study. LVEF at least 50%; Controlled blood glucose if diabetic; controlled Blood pressure if hypertensive
* Pulmonary: No severe pulmonary disease that would limit normal life expectancy or preclude study
* Others: HIV negative status; No prior haematological cancers or chemotherapy or radiation therapy in the past

Exclusion Criteria:

* Pregnancy
* Nursing mothers

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of interim PET guided therapy strategy interms of EFS in advanced HL | Once in a year
  This is a phase II design looking at the efficacy of response adapted therapy delivering Esc BEACOPP in select patients with positive interim PET CT while PET negative patients continue to receive ABVD

SECONDARY OUTCOMES:
Toxicity of escalated BEACOPP | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prasanth Ganesan, MD, DM, Principal Investigator — Cancer Institute (WIA) , Adyar, Chennai
Locations (1):
- Department of Medical Oncology, Cancer Institute (WIA), Adyar, Chennai, Tamil Nadu, India

REFERENCES:
- [Derived] Ganesan P, Rajendranath R, Kannan K, Radhakrishnan V, Ganesan TS, Udupa K, Lakshmipathy KM, Mahajan V, Sundersingh S, Rajaraman S, Krishnakumar R, Sagar TG. Phase II study of interim PET-CT-guided response-adapted therapy in advanced Hodgkin's lymphoma. Ann Oncol. 2015 Jun;26(6):1170-1174. doi: 10.1093/annonc/mdv077. Epub 2015 Feb 20. PMID 25701453